CLINICAL TRIAL: NCT02556489
Title: Transcriptomics Signature of Anti Vaccinia Memory B Cells in Healthy Individuals at a Short Time After Vaccination
Brief Title: Transcriptomics Signature of Anti Vaccinia Memory B Cells
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C15-23; 2015-A00752-47 (Registry Identifier: IDRCB)
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-05

CONDITIONS: Healthy
Keywords: immunological memory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Analyse the transcriptomic signature of anti vaccinia memory B cells at a short time after vaccination as compared to the signature already established in long-lived memory B cells.

ELIGIBILITY:
Inclusion Criteria:

* Healthy donors vaccinated against smallpox

Exclusion Criteria:

* none

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy donnors vaccinated against smallpox
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
signature of anti vaccinia long-lived memory B cells | 12 months